CLINICAL TRIAL: NCT03379662
Title: A Double-blind, Placebo-controlled Randomized Evaluation of the Effect of the Erchonia® HLS Laser Device on Children and Adolescents With Autistic Disorder
Brief Title: An Evaluation of Low Level Laser Light Therapy for Autistic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC_AUT_001
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Autistic Disorder
Keywords: Autism; Autistic Disorder; Autistic Spectrum Disorder; Irritability; laser; light therapy
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Erchonia HLS Laser (Experimental): The Erchonia HLS Laser is administered 8 times across 4 weeks for 5 minutes each time to the skull at the base of the brain and temporal areas.
  Interventions: Device: Erchonia HLS Laser
- Placebo Laser (Placebo Comparator): The Placebo Laser is administered 8 times across 4 weeks for 5 minutes each time to the skull at the base of the brain and temporal areas.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia HLS Laser — The Erchonia HLS Laser emits a 640 nm (nanometer) wavelength with a tolerance of ±10 nm from each of two 7.5 mw (milliwatt) laser diodes.
  Arms: Erchonia HLS Laser
Device: Placebo Laser — The Placebo Laser emit the same visible light output as the active HLS Laser but without therapeutic effect.
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether the Erchonia HLS Laser is effective in the treatment of irritability associated with autistic disorder in children and adolescents aged five (5) to seventeen (17) years.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a range of complex neurodevelopment disorders characterized by behavioral, developmental, cognitive and psychological deficits that include social impairment, communication and language difficulties, hyperactivity, irritability, obsessive interests and restricted, and repetitive behaviors. Autistic disorder, sometimes called autism or classical ASD, is the most severe form of ASD. ASD occurs in all ethnic and socioeconomic groups and affects every age group, with symptoms appearing before age 3. The Centers for Disease Control (CDC) estimates that 1 out of 88 children age 8 will have an ASD, with males four times more likely to have an ASD than females.

There is no cure for ASD and no single best treatment for all individuals with autistic disorder. The majority of diagnosed cases of autism are idiopathic with an enigmatic pathogenesis, and as a result, therapeutic approaches have focused on mitigating specific symptoms rather than treating disease etiologies. The current standard treatment approach is a team approach to customize an individual highly structured, specialized program or treatment plan including medications, therapies and behavioral interventions targeted toward improving the individual's specific symptoms.

The cause of ASD is not clearly understood, but it is believed that both genetics and environment likely play a role. Magnetic resonance imaging (MRI) studies have demonstrated increased brain volume and head circumference during early developmental childhood, suggesting that autistic brains experience a period a rapid overgrowth which hampers further development during later developmental stages. Morphological aberrations have been observed in the hippocampus, anterior cingulate cortex, prefrontal cortex, amygdala, and cerebellum. Another consistent observation has also been the reduction in cerebellar vermis volume, which helps to explain specific behavioral patterns in children.

Molecular analysis of postmortem brain tissue has revealed reduced Purkinje cell numbers, which helps to explain aberrant locomotive activity and level presser function. Another finding has been impaired neuronal connectivity within the cerebellum, amygdala, anterior cingulate cortex, and dorsolateral prefrontal cortex. As a consequence, synapse structure and function has demonstrated impairment in postmortem evaluations. Dendritic spines of glutamatergic neurons in autistic patients have shown morphological alterations and suppressed density, which, in turn, results in diminished synaptic transmissions. Nascent spines have been reported in frontal, temporal, and parietal cortices of autistic patients, and have a negative correlation with cognitive abilities in autism. Other neurological aberrations include signaling through metabotropic glutamate receptor (mGluR) and ƴ-aminobutyric acid (GABA)ergic system.

The elusive pathophysiology of autism provides a marked challenge for health care providers. One promising technology is low-level laser therapy (LLLT). LLLT uses photonic energy to modulate the behavior and function of cells by stimulating molecular entities capable of absorbing discrete wavelengths. or instance, cytochrome c oxidase (CCO), a terminal enzyme of the respiratory change, contains a tetrapyrrole prosthetic group that has been shown to absorb 635nm. Photon-induced activation of CCO increases cell bioenergetics, which, in turn, activates intra-cellular secondary signaling cascades that in turn affect growth factor synthesis, cell proliferation, cytokine production, and expression of specific transcription factors. Studies have reported increased adenosine triphosphate (ATP) synthesis along with activation of the intracellular redox state following the production of reactive oxygen species (ROS). As an essential bio-catalyst, ATP lowers the activation for pivotal biochemical reactions within cells. Concerning neurons, laser irradiation has been shown to promote the recovery of injured peripheral nerves and the spinal cord. Moreover, studies have revealed that excitable cells like neurons can be directly stimulated by light, enhancing the action potential of the cell increasing the release of neurotransmitters such as glutamate and acetylcholine.

Clinical outcomes with LLLT trials include nerve regeneration, increased neurotransmitter release, growth factor synthesis, and neovascularization to name a few. It follows that positioning of the laser along impaired regions of an autistic brain could elicit a positive therapeutic outcome in a safe and non-invasive manner.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child or adolescent aged 5 to 17 years
* Meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision criteria (DSM-IV-TR) for autistic disorder within the past 2 years, as diagnosed by a trained, qualified medical professional such as a pediatric neurologist, child psychiatrist or developmental pediatrician
* Diagnosis is confirmed by Autism Diagnostic Interview (ADI-R)
* Demonstrates 'irritable' behaviors such as tantrums, aggression, self-injurious behavior, or a combination of such behaviors
* Aberrant Behavior Checklist (ABC) Irritability Subscale score is >=18
* Clinical Global Impressions - Severity (CGI-S) scale score is >=4 (moderately ill)
* Current therapeutic/intervention plan for treating autistic disorder has been consistent/ stable over at least the past 3 months
* Caregiver agrees, and it is possible for, the subject to abstain from partaking in new treatments to treat autistic disorder symptoms during the course of study participation
* Female subjects of child-bearing age are willing and able to use acceptable means of contraception throughout study participation.

Exclusion Criteria:

* Primary or concurrent diagnosis of another disorder or other identifiable genetic condition associated with the autism spectrum scale or with mental retardation, including:

Pervasive Developmental Disorder-Not Otherwise Specified (PDD-NOS); Asperger's Disorder; Rett's Disorder; Fragile-X Syndrome; Childhood Disintegrative Disorder; Down Syndrome

* Seizure disorders (active), cerebrovascular disease or brain trauma as etiology of autistic behavior
* Current diagnosis of, and treatment for, bipolar disorder, psychosis, schizophrenia, or major depression
* Current use of a psychotropic drug deemed effective for the treatment of aggression, tantrums or self-injurious behavior
* Known neurological disease, such as encephalitis
* Significant sensory or motor impairment such as cerebral palsy
* Diagnosis of epilepsy that is currently treated with anti-convulsant medication
* Previous significant head trauma
* Hearing loss requiring use of assistive devices such as hearing aids or cochlear implant
* Significant visual impairment that cannot be adequately corrected with lenses
* Documented mental age younger than 18 months
* HIV and other autoimmune disorders
* Active cancer or treatment for cancer within last 6 months
* Unstable cardiac disease, such as a recent cardiac arrhythmias (including atrial fibrillation, ventricular fibrillation and irregular atrial-ventricular conduction time), or recent congestive heart failure, or recent myocardial infarction
* Previous surgical interventions to the head/neck area
* Sensitivity to, or contraindication for, light therapy
* Subject is presently pregnant or breast feeding
* Participation in a research study within the past 30 days

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calixto Machado, MD, Principal Investigator
Locations (1):
- Institute for Brain and Rehabilitation Sciences, Nazareth, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia HLS Laser | Placebo Laser
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia HLS Laser | Placebo Laser | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.24 (3.02) | 8.37 (3.15) | 8.29 (3.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 12 | 20
  White | 12 | 4 | 16
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Cuba | 21 | 19 | 40
Baseline Aberrant Behavior Checklist (ABC) Irritability Score [Mean (Standard Deviation); unit: score on a scale] — The ABC Irritability Subscale includes questions about aggression, self-injury, tantrums, agitation and unstable mood on a scale of 0 to 45, with higher scores indicating greater severity. Data from studies of developmentally disabled children indicated that a score of 18 is 1.3 to 1.5 SD above the population means, depending on the age and sex of the child.
  score on a scale | 30.52 (15.71) | 29.58 (28.89) | 30.04 (22.65)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Study Endpoint in the Aberrant Behavior Checklist (ABC) Irritability & Agitation Subscale Score.
Description: Primary outcome measure in this study is defined as the mean change from baseline to 4 weeks of intervention (study endpoint), in the Aberrant Behavior Checklist (ABC) Irritability Subscale score. The ABC Irritability Subscale contains 15 items relating to aggression, self-injury, tantrums, agitation and unstable mood in individuals with developmental disorders. Each item is rated from 0 (not at all a problem) to 3 (the problem is severe in degree). The individual scores are summed for a total score from 0 to 45, with higher scores indicating greater severity. A negative (-) change indicates a decrease in symptom severity and is positive for improvement. A positive (+) change indicates an increase in symptom severity and is negative for improvement. Study success is established as the detection of a minimum mean difference of -8.5 points between test and placebo groups in the change in ABC Irritability Subscale score.
Time Frame: Baseline and 4 weeks (Study Endpoint)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erchonia HLS Laser | Placebo Laser
Number analyzed (Participants) | 21 | 19
score on a scale | -14.81 (6.40) | 0.37 (1.38)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Erchonia HLS Laser | Placebo Laser
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-01-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT03379662/Prot_SAP_ICF_000.pdf